CLINICAL TRIAL: NCT06066554
Title: Assessment of the Tissue and Serum Level of NLRP1, NLRP3 Inflammasomes and Interleukin-18 in Early Stages of Mycosis Fungoids Patients Before and After Different Treatment Modalities: Controlled Clinical Trial.
Brief Title: Tissue and Serum Level of NLRP1, NLRP3 and Il-18 in Early Stages of mf Patients
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Nourhan Emad, Assistant lecturer, Cairo University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: MD_437_2022
Record Dates: First submitted 2023-09-27; First posted 2023-10-04 (Actual); Last update posted 2024-02-06 (Actual); Status verified 2024-02

CONDITIONS: Early Disease Onset
MeSH Terms: interventions — Photochemotherapy

STUDY DESIGN:
Intervention Model Description: Thirty new patients with early stage mycosis fungoids will be allocated to proper treatment modality that differ according to the patient's clinical state following kasralainy phototherapy unit protocol
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- 14 early mycosis fungoids patients (Active Comparator): Puva (psoralin and uva) Measure nlrp1 and nlrp3 and il18
  Interventions: Device: Puva (psoralin and uva )
- 8 mycosis fungoids patients (Active Comparator): Puva (psoralin and uva) and methotrexate Measure nlrp1 and nlrp3 and il18
  Interventions: Device: Puva (psoralin and uva )
- Eight mycosis fungoids patients (Active Comparator): Puva (psoralin and uva)and retinoids (acetritin) Measure nlrp1 and nlrp3 and il18
  Interventions: Device: Puva (psoralin and uva )
- Controls (No Intervention): Measure nlrp1 and nlrp3 and il18

INTERVENTIONS:
Device: Puva (psoralin and uva ) — Intervention will be given for 48 sessions or till coplete resolution of biopsied plaque
  Other Names: Methotrexate; Retinoids
  Arms: 14 early mycosis fungoids patients; 8 mycosis fungoids patients; Eight mycosis fungoids patients

SUMMARY:
To compare tissue and serum level of NLRP1, NLRP3 inflammasomes and Interleukin (IL)-18 in mycosis fungoids patients and normal controls.

To compare tissue and serum level of NLRP1, NLRP3 inflammasomes and Interleukin (IL)-18 in mycosis fungoids patients before and after different treatment modalities.

DETAILED DESCRIPTION:
Thirty patients with early stage mycosis fungoids and thirty normal healthy controls will be recruited. An informed written consent will be obtained from all patients and controls.

Data collection Demographic data Each patient will be subjected to detailed history taking as regards age, sex, residence, marital status, smoking, special habits of medical importance, duration of the disease, associated diseases, previous therapy and family history.

Evaluation of the clinical response The patients will be photographed and evaluated at baseline and at the end of treatment .

Clinical scoring of five mycosis fungoids skin lesions will be done using Composite assessment of index lesion severity (CAILS) (Oslen et al., 2011).

Clinical scoring of whole body affection will be done using Modified Severity Weighted Assessment tool (MSWAT) (Oslen et al., 2011).

Assessment of response of mycosis fungoids patients to our treatment modalities will be done using Objective response rate (ORR) (Oslen et al., 2011).

Treatment (therapeutic intervention):

Thirty new patients with early stage mycosis fungoids will be allocated to proper treatment modality that differ according to the patient's clinical state following kasralainy phototherapy unit protocol End of the study will be defined as achieving clinically near complete clearance of the lesion from which a tissue biopsy will be taken or a maximum of 48 sessions of treatment.

Biochemical assessment and pathological assessment (Diagnostic intervention) :

Two lesional skin 4 mm punch biopsies will be taken from same lesion in all thirty patients and once from all thirty normal healthy controls.

Three milliliter serum samples will be taken from all thirty patient before and after treatment and once from all thirty healthy controls.

one skin biopsy and serum samples before treatment will be subjected to biochemical assessment for measurement of NLRP1, NLRP3 inflammasomes and Interleukin (IL)-18 by ELISA (Enzyme linked immunosorbent assay) technique.

The other skin biopsy will be used for pathological assessment. The same process will be repeated after treatment for patients only to assess the percent change in all parameters and in lymphocytic infiltration .

Fate of tissue and serum samples Tissue samples used for biochemical assessment will be completely crushed to extract protein for ELISA, any residual biological tissue will be safely discarded in the incinerator.

Tissue samples used for pathological assessment will be put on paraffin blocks then on slides that will be kept in our department.

Serum samples will be collected in special containers to be sent to the official site in the hospital to get rid of them.

Intervention:

Diagnostic intervention : biochemical assessment for measurement of NLRP1, NLRP3 inflammasomes and Interleukin (IL)-18 by ELISA (Enzyme linked immunosorbent assay) technique in tissue and serum samples of all thirty patients and healthy controls.

Therapeutic intervention : Thirty new patients with early stage mycosis fungoids will be allocated to proper treatment modality that differ according to the patient's clinical state following kasralainy phototherapy unit protocol

ELIGIBILITY:
Inclusion Criteria:

* New patients with early stages of mycosis fungoids (patch and plaque stage).
* Both genders
* Age group ≥ 18 years old.

Exclusion Criteria:

* Patients with late stages mycosis fungoids (Tumor stage).
* Patients with absolute contraindication to phototherapy (e.g. any other skin cancers or photosensitivity); or to psoralen (e.g. liver disease).
* Subjects with history of solid or hematological malignancy as leukemia.
* Patients with autoimmune disease (e.g. SLE).
* Patients who received treatment of mycosis fungoids for the past one month.
* Pregnant and lactating females.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-02-15 (Estimated); Primary Completion 2024-05-15 (Estimated); Study Completion 2024-05-30 (Estimated)

PRIMARY OUTCOMES:
To compare tissue and serum level of NLRP1, NLRP3 inflammasomes and Interleukin (IL)-18 in mycosis fungoids patients and normal controls. | 4 months
  Diagnostic

SECONDARY OUTCOMES:
To compare tissue and serum level of NLRP1, NLRP3 inflammasomes and Interleukin (IL)-18 in mycosis fungoids patients before and after different treatment modalities. | 4 months
  Intervention of 48 sessions of puva alone or in addition to mtx or retinoids
Correlating tissue and serum level of NLRP1, NLRP3 inflammasomes and Interleukin (IL)-18 in mycosis fungoids patients with patient's age, sex, duration of disease, extent of disease. | 4 months
  Observational

IPD SHARING:
Plan to Share IPD: Yes
Data will be shared after paper submission
Supporting Information: Study Protocol
Time Frame: Around 4 months
Access Criteria: nourhanemad921@gmail.com